CLINICAL TRIAL: NCT02282293
Title: Reducing the Burden of Malaria in HIV-Infected Pregnant Women and Their HIV-Exposed Children (PROMOTE Birth Cohort 2)
Brief Title: Reducing the Burden of Malaria in HIV-Infected Pregnant Women and Their HIV-Exposed Children (PROMOTE-BC2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Diana Havlir, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROMOTE-BC2
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Malaria; Human Immunodeficiency Virus
Keywords: Chemoprevention; Malaria; Uganda; Dihydroartemisinin-piperaquine; Trimethoprim-sulfamethoxazole; Human Immunodeficiency Virus
MeSH Terms: conditions — Malaria; Acquired Immunodeficiency Syndrome | interventions — Sulfamethoxazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daily TS + Monthly DP pregnancy (Active Comparator): Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) every 4 weeks during pregnancy. During pregancy, TS will be given to women at a dose of 960mg once daily.
  Interventions: Drug: Monthly dihydroartemisinin-piperaquine (DP) + daily trimethoprim/sulfamethoxazole (TS)
- Daily TS + DP Placebo pregnancy (Placebo Comparator): Women will be given DP placebo (3 tabs, given once a day for 3 consecutive days) every 4 weeks during pregnancy. During pregnancy, TS will be given to women at a dose of 960mg once daily.
  Interventions: Drug: Monthly placebo + daily trimethoprim/sulfamethoxazole (TS)

INTERVENTIONS:
Drug: Monthly dihydroartemisinin-piperaquine (DP) + daily trimethoprim/sulfamethoxazole (TS)
  Other Names: Duo-Cotexin (Holley-Cotec)
  Arms: Daily TS + Monthly DP pregnancy
Drug: Monthly placebo + daily trimethoprim/sulfamethoxazole (TS)
  Arms: Daily TS + DP Placebo pregnancy

SUMMARY:
This is a double-blinded, randomized controlled trial of 200 HIV-infected pregnant women living in Tororo, Uganda, an area of high malaria transmission. HIV-infected pregnant women between 12 and 28 weeks gestation will be randomized to receive enhanced malaria chemoprevention with monthly dihydroartemisinin-piperaquine (DP) versus monthly DP placebo. Their HIV-exposed children will receive the same prevention regimen from 2 to 24 months of age to which the mothers were randomized. All women will receive daily trimethoprim-sulfamethoxazole (TS) throughout the study per Uganda Ministry of Health guidelines. Children will also receive daily TS from 6 weeks to 24 months of age. TS will be considered a study drug only in infants and children beginning 6 weeks after cessation of breastfeeding and upon exclusion of HIV infection. Women and their children will be followed for 36 months after delivery. In a subset of the study population, the investigators will conduct an intensive pharmacokinetic study that will evaluate pharmacokinetic exposure of DP and EFV. The investigators will also measure HIV-related outcomes among the women enrolled in the study. The investigators will test the hypothesis that for HIV-infected mothers and HIV-exposed infants, that enhanced versus standard malaria chemoprevention in HIV-infected pregnant women and their children will reduce the incidence of malaria among children from 0 to 24 months of age and improve the development of naturally acquired antimalarial immunity.

DETAILED DESCRIPTION:
Pregnant women will be scheduled to be seen in the study clinic every 4 weeks during their pregnancy. Women will be seen at 1 week, 6 weeks, and 3 months postpartum and every 3 months thereafter. In addition, pregnant women will be instructed to come to the study clinic for all their medical care and avoid the use of any outside medications. Women will be provided all routine HIV care at the clinic according to Uganda MOH guidelines. All women will have ARVs and TS dispensed at the study clinic. Counseling on breastfeeding and infant feeding will be provided per Uganda MOH guidelines. HIV care and breastfeeding and infant feeding recommendations may be changed to reflect the most recent standard of care per MOH guidelines. Children will be scheduled to be seen in the clinic every 4 weeks and parents /guardians of children will be instructed to bring their child to the study clinic for all medical care and avoid the use of any outside medications. The study clinic will remain open 7 days a week from 8 a.m. to 5 p.m.

Each time a study participant is seen in the clinic a standardized history and physical exam will be performed. Patients who are febrile (tympanic temperature > 3 8.0˚C) or report history of fever in the past 24 hours will have blood obtained by finger prick for a thick blood smear. If the thick blood smear is positive, the patient will be diagnosed with malaria. If the thick blood smear is negative, the patient will be managed by study physicians for a non-malarial febrile illness. If the patient is afebrile and does not report a recent fever, a thick blood smear will not be obtained, except when following routine testing schedules.

Routine assessments will be done in the clinic every 4 weeks for both pregnant women and children. Pregnant women and children will receive standards of care as designated in the Uganda MOH guidelines. Children will have care for HIV-exposed children according to MOH guidelines, with the exception that TS will be continued until 2 years of life. Routine care in children will use Integrated Management of Childhood Illness (IMCI) guidelines. During routine assessments subjects will be asked about visits to outside health facilities and the use of any medications outside the study protocol. Standardized assessment of adherence will also be done for study drugs administered at home and Insecticide Treated Net use. A routine history and physical exam will be performed using a standardized clinical assessment form. Blood will be collected by finger prick for thick smear, collection of plasma for PK studies, and filter paper samples. Phlebotomy for routine laboratory tests (CBC and ALT) to monitor for potential adverse events from study medications and for immunology studies will be performed every 8 weeks in pregnant women. Non malaria screening will also include stool ova and parasite examination, circulating filarial antigens (by ICT card for Wucheria), and blood smear for microfilaremia (including Mansonella perstans) using Knott's technique. For pregnant women, study drugs will be administered at the time of each routine visit.

ELIGIBILITY:
Inclusion Criteria:

1. Intrauterine pregnancy confirmed by ultrasound
2. Estimated gestational age between 12-28 weeks
3. Confirmed to be HIV-infected by Uganda country standard rapid HIV test
4. 16 years of age or older
5. Residency within 30 km of the study clinic
6. Provision of informed consent
7. Agreement to come to the study clinic for any febrile episode or other illness and avoid medications given outside the study protocol
8. Plan to deliver in the hospital

Exclusion Criteria:

1. History of serious adverse event to TS or DP
2. Refusal to take cART during pregnancy or as part of routine HIV care
3. Active medical problem requiring inpatient evaluation at the time of screening
4. Intention of moving more than 30 km from the study clinic
5. Active WHO stage 4 condition not stable under treatment
6. Signs or symptoms of early or active labor
7. Currently on ritonavir
8. Currently taking drugs associated with known risk of Torsades de pointes
9. Currently taking CYP3A inhibitor medications which potentially inhibit the metabolism of piperaquine
10. History of cardiac problems or fainting

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane V Havlir, MD, Principal Investigator — University of California, San Francisco; Grant Dorsey, MD, PhD, Principal Investigator — University of California, San Francisco; Moses R Kamya, MBChB, MMed, PhD, Principal Investigator — Makerere University; Infectious Diseases Research Collaboration
Locations (1):
- IDRC Research Clinic - Tororo District Hospital, Tororo, Uganda

REFERENCES:
- [Background] Kajubi R, Huang L, Jagannathan P, Chamankhah N, Were M, Ruel T, Koss CA, Kakuru A, Mwebaza N, Kamya M, Havlir D, Dorsey G, Rosenthal PJ, Aweeka FT. Antiretroviral Therapy With Efavirenz Accentuates Pregnancy-Associated Reduction of Dihydroartemisinin-Piperaquine Exposure During Malaria Chemoprevention. Clin Pharmacol Ther. 2017 Sep;102(3):520-528. doi: 10.1002/cpt.664. Epub 2017 May 30. PMID 28187497
- [Background] Sonoiki E, Nsanzabana C, Legac J, Sindhe KM, DeRisi J, Rosenthal PJ. Altered Plasmodium falciparum Sensitivity to the Antiretroviral Protease Inhibitor Lopinavir Associated with Polymorphisms in pfmdr1. Antimicrob Agents Chemother. 2016 Dec 27;61(1):e01949-16. doi: 10.1128/AAC.01949-16. Print 2017 Jan. PMID 27821443
- [Result] Natureeba P, Kakuru A, Muhindo M, Ochieng T, Ategeka J, Koss CA, Plenty A, Charlebois ED, Clark TD, Nzarubara B, Nakalembe M, Cohan D, Rizzuto G, Muehlenbachs A, Ruel T, Jagannathan P, Havlir DV, Kamya MR, Dorsey G. Intermittent Preventive Treatment With Dihydroartemisinin-Piperaquine for the Prevention of Malaria Among HIV-Infected Pregnant Women. J Infect Dis. 2017 Jul 1;216(1):29-35. doi: 10.1093/infdis/jix110. PMID 28329368
- [Result] Prahl M, Jagannathan P, McIntyre TI, Auma A, Wamala S, Nalubega M, Musinguzi K, Naluwu K, Sikyoma E, Budker R, Odorizzi P, Kakuru A, Havlir DV, Kamya MR, Dorsey G, Feeney ME. Sex Disparity in Cord Blood FoxP3+ CD4 T Regulatory Cells in Infants Exposed to Malaria In Utero. Open Forum Infect Dis. 2017 Feb 11;4(1):ofx022. doi: 10.1093/ofid/ofx022. eCollection 2017 Winter. PMID 28480292
- [Result] Odorizzi PM, Feeney ME. Impact of In Utero Exposure to Malaria on Fetal T Cell Immunity. Trends Mol Med. 2016 Oct;22(10):877-888. doi: 10.1016/j.molmed.2016.08.005. Epub 2016 Sep 7. PMID 27614925
- [Result] Prahl M, Jagannathan P, McIntyre TI, Auma A, Farrington L, Wamala S, Nalubega M, Musinguzi K, Naluwu K, Sikyoma E, Budker R, Vance H, Odorizzi P, Nayebare P, Ategeka J, Kakuru A, Havlir DV, Kamya MR, Dorsey G, Feeney ME. Timing of in utero malaria exposure influences fetal CD4 T cell regulatory versus effector differentiation. Malar J. 2016 Oct 7;15(1):497. doi: 10.1186/s12936-016-1545-6. PMID 27717402
- [Result] Roh ME, Shiboski S, Natureeba P, Kakuru A, Muhindo M, Ochieng T, Plenty A, Koss CA, Clark TD, Awori P, Nakalambe M, Cohan D, Jagannathan P, Gosling R, Havlir DV, Kamya MR, Dorsey G. Protective Effect of Indoor Residual Spraying of Insecticide on Preterm Birth Among Pregnant Women With HIV Infection in Uganda: A Secondary Data Analysis. J Infect Dis. 2017 Dec 19;216(12):1541-1549. doi: 10.1093/infdis/jix533. PMID 29029337
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Hughes E, Imperial M, Wallender E, Kajubi R, Huang L, Jagannathan P, Zhang N, Kakuru A, Natureeba P, Mwima MW, Muhindo M, Mwebaza N, Clark TD, Opira B, Nakalembe M, Havlir D, Kamya M, Rosenthal PJ, Dorsey G, Aweeka F, Savic RM. Piperaquine Exposure Is Altered by Pregnancy, HIV, and Nutritional Status in Ugandan Women. Antimicrob Agents Chemother. 2020 Nov 17;64(12):e01013-20. doi: 10.1128/AAC.01013-20. Print 2020 Nov 17. PMID 33020153
- [Derived] Wallender E, Zhang N, Conrad M, Kakuru A, Muhindo M, Tumwebaze P, Kajubi R, Mota D, Legac J, Jagannathan P, Havlir D, Kamya M, Dorsey G, Aweeka F, Rosenthal PJ, Savic RM. Modeling Prevention of Malaria and Selection of Drug Resistance with Different Dosing Schedules of Dihydroartemisinin-Piperaquine Preventive Therapy during Pregnancy in Uganda. Antimicrob Agents Chemother. 2019 Jan 29;63(2):e01393-18. doi: 10.1128/AAC.01393-18. Print 2019 Feb. PMID 30530597
- [Derived] Wallender E, Vucicevic K, Jagannathan P, Huang L, Natureeba P, Kakuru A, Muhindo M, Nakalembe M, Havlir D, Kamya M, Aweeka F, Dorsey G, Rosenthal PJ, Savic RM. Predicting Optimal Dihydroartemisinin-Piperaquine Regimens to Prevent Malaria During Pregnancy for Human Immunodeficiency Virus-Infected Women Receiving Efavirenz. J Infect Dis. 2018 Mar 5;217(6):964-972. doi: 10.1093/infdis/jix660. PMID 29272443

RESULTS

PARTICIPANT FLOW:
Groups:
- TS + DP Placebo Pregnancy: Women will be given DP placebo (3 tabs, given once a day for 3 consecutive days) every 4 weeks during pregnancy. During pregnancy, TS will be given to women at a dose of 960mg once daily.
  Infants will be given DP placebo (tablets once a day for 3 consecutive days) every four weeks from 2 months to 24 months of age. Infants will be given TS daily starting at 6 weeks of life using weight-based guidelines.
  Placebo
- Daily TS + Monthly DP Pregnancy: Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) every 4 weeks during pregnancy. During pregancy, TS will be given to women at a dose of 960mg once daily.
  Infants will be given DP (half strength tablets once a day for 3 consecutive days) every four weeks from 2 months to 24 months of age. Infants will be given TS daily starting at 6 weeks of life using weight-based guidelines.
  Monthly dihydroartemisinin-piperaquine (DP) for adult women during pregnancy
  Monthly dihydroartemisinin-piperaquine (DP) for infants
Period: Overall Study
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy
Started | 100 | 100
Completed | 97 | 97
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Unable to comply with study procedures | 1 | 0
Not completed — Moved out of study area | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (5.8) | 29.8 (6.8) | 30.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 100 | 100 | 200
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Gestational age (cont) [Mean (Standard Deviation); unit: weeks] | 19.2 (4.1) | 19.9 (4.5) | 19.6 (4.3)
Gestational age (cat) [Count of Participants; unit: Participants]
  12-16 wk | 28 | 25 | 53
  > 16-20 wk | 30 | 26 | 56
  > 20 - 24 wk | 29 | 27 | 56
  > 24 - 28 wk | 13 | 22 | 35
Gravidity [Count of Participants; unit: Participants]
  1 pregnancy | 5 | 13 | 18
  2 pregnancy | 13 | 12 | 25
  >= 3 pregnancies | 82 | 75 | 157
Insecticide-treated bednet (ITN) ownership [Count of Participants; unit: Participants] | 57 | 57 | 114
Household Wealth [Count of Participants; unit: Participants]
  Lowest Tertile | 33 | 34 | 67
  Middle Tertile | 30 | 36 | 66
  Highest Tertile | 37 | 30 | 67
Receiving TMP-SMX prophylaxis [Count of Participants; unit: Participants] | 90 | 91 | 181
Receiving ART [Count of Participants; unit: Participants] | 82 | 79 | 161
CD4+ T-cell count, cells/mm^3 [Median (Inter-Quartile Range); unit: cells/mm^3] | 500 [392 to 622] | 516 [368 to 660] | 516 [372 to 638]
HIV load below limit of detection [Count of Participants; unit: Participants] | 51 | 60 | 111
WHO HIV disease stage [Count of Participants; unit: Participants] — WHO clinical staging of HIV/AIDS is defined in the following document: https://www.who.int/hiv/pub/guidelines/clinicalstaging.pdf
  In brief:
  Stage 1. Asymptomatic Stage 2. Minor infections or <10% weight loss Stage 3. TB, bacterial infections; systemic symptoms or laboratory values of chronic illness Stage 4. Opportunistic infections or cancers
  Participants
    WHO Stage 1 | 93 | 97 | 190
    WHO Stage 2 | 4 | 1 | 5
    WHO Stage 3 | 3 | 2 | 5
    WHO Stage 4 | 0 | 0 | 0
Detection of malaria parasites by LAMP [Count of Participants; unit: Participants] | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Placental Malaria
Description: The primary outcome will be the prevalence of placental malaria based on placental histopathology and dichotomized into any evidence of placental infection (parasites or pigment) vs. no evidence of placental infection.
Time Frame: at delivery estimated to be within 10 to 30 weeks of study entry
Measure: Count of Participants; unit: Participants
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy
Number analyzed (Participants) | 96 | 98
Participants | 3 | 6
Statistical Analysis 1: Comparison: TS + DP Placebo Pregnancy vs Daily TS + Monthly DP Pregnancy; Test type: Other; p = 0.50, Chi-squared — Calculated p-value; Risk Ratio (RR) = 1.96, 95% CI 2-sided [0.50 to 7.61]

2. Primary Outcome: Incidence of Malaria, Pregnant Women
Description: The primary outcome will be the incidence of malaria, defined as the number of incident episodes per time at risk. Incident cases will include all treatments for malaria not proceeded by another treatment in the previous 14 days.
Time Frame: Time at risk will begin following administration of first dose of study drug to delivery
Measure: Number; unit: Events per person-year
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy
Number analyzed (Participants) | 100 | 100
Events per person-year | 0.03 | 0.00

3. Secondary Outcome: Maternal Parasitemia at Delivery by Microscopy and LAMP
Description: Proportion of women with parasitemia detected by microscopy or LAMP at delivery
Time Frame: At delivery
Population: Out of all 100 enrolled women in each arm: two women in TS+Placebo arm did not have maternal blood specimens collected to analyze; One participant in Daily TS + Monthly DP pregnancy arm did not have blood slide completed for microscopy results but did have blood spot collected for LAMP analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy
Number analyzed (Participants) | 98 | 100
Participants
  Microscopy: number analyzed (Participants) | 98 | 99
  Microscopy | 0 | 1
  LAMP | 2 | 4
Statistical Analysis 1: Comparison: TS + DP Placebo Pregnancy vs Daily TS + Monthly DP Pregnancy; Test type: Other; p = 0.50, Chi-squared; Risk Ratio (RR) = 1.96, 95% CI 2-sided [0.50 to 7.61]

4. Secondary Outcome: Placental Parasitemia (Number of Women With Placental Blood Samples Positive for Malaria by Microscopy or PCR)
Description: Proportion of placental blood samples positive for malaria by microscopy or PCR
Time Frame: At delivery
Population: Out of all 100 enrolled women in each arm: four women in TS+Placebo arm and two women in TS+DP arm did not have placental blood specimens collected to analyze; One participant TS+Placebo arm did not have microscopy results; Only one placental blood specimen was collected for each woman
Measure: Count of Participants; unit: Participants
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy
Number analyzed (Participants) | 96 | 98
Participants
  Microscopy of placental blood: number analyzed (Participants) | 95 | 98
  Microscopy of placental blood | 0 | 1
  LAMP analysis of placental blood | 1 | 3

5. Secondary Outcome: Number of Monthly Routine Visits With Positive Blood Samples for Parasites
Description: Proportion of monthly routine blood samples positive by LAMP for parasites
Time Frame: Following administration of first dose of study drug to delivery
Measure: Count of Units; unit: visits with positive blood sample
Units Other Than Participants: visits with positive blood sample
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy
Number analyzed (Participants) | 100 | 100
Number analyzed (visits with positive blood sample) | 392 | 368
visits with positive blood sample | 12 | 5
Statistical Analysis 1: Comparison: TS + DP Placebo Pregnancy vs Daily TS + Monthly DP Pregnancy; Test type: Other; p = 0.19, GEE — Calculated p-value; Risk Ratio (RR) = 0.45, 95% CI 2-sided [0.13 to 1.48]

6. Secondary Outcome: Composite Adverse Birth Outcome (Proportion With Low Birth Weight (<2500 gm), Spontaneous Abortion (<28 Weeks), Stillbirth (Fetal Demise ≥28 Weeks), Congenital Anomaly, or Preterm Delivery (<37 Weeks)
Description: Proportion with low birth weight (<2500 gm), spontaneous abortion (<28 weeks), stillbirth (fetal demise ≥28 weeks), congenital anomaly, or preterm delivery (<37 weeks)
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy
Number analyzed (Participants) | 100 | 100
Participants | 15 | 20
Statistical Analysis 1: Comparison: TS + DP Placebo Pregnancy vs Daily TS + Monthly DP Pregnancy; Test type: Other; p = 0.35, Chi-squared; Risk Ratio (RR) = 1.33, 95% CI 2-sided [0.72 to 2.45]

7. Secondary Outcome: Number of Routine Visits Measured Every 8 Weeks During Pregnancy for Which the Participants Had Anemia
Description: Anemia (hemoglobin less than 11g/dL) measured every 8 weeks during pregnancy
Time Frame: Following administration of first dose of study drugs to delivery
Measure: Count of Units; unit: Routine visit done every 8 weeks
Units Other Than Participants: Routine visit done every 8 weeks
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy
Number analyzed (Participants) | 100 | 100
Number analyzed (Routine visit done every 8 weeks) | 206 | 191
Routine visit done every 8 weeks | 65 | 51

ADVERSE EVENTS:
Time Frame: Following administration of first study drug to 6 weeks postpartum
Arm/Group | TS + DP Placebo Pregnancy | Daily TS + Monthly DP Pregnancy
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 4/100 | 6/100
Other Adverse Events (participants affected / at risk) | 92/100 | 91/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TS + DP Placebo Pregnancy (N=100) | Daily TS + Monthly DP Pregnancy (N=100)
Anemia (Blood and lymphatic system disorders) | 3 | 2
Congenital anomaly (Congenital, familial and genetic disorders) | 1 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TS + DP Placebo Pregnancy (N=100) | Daily TS + Monthly DP Pregnancy (N=100)
Abdominal pain (General disorders) | 68 (85) | 63 (74)
Cough (General disorders) | 41 (69) | 43 (55)
Headache (General disorders) | 34 (39) | 37 (43)
Anemia (Blood and lymphatic system disorders) | 40 (49) | 38 (45)
Malaise (General disorders) | 24 (27) | 21 (24)
Diarrhea (General disorders) | 14 (17) | 11 (14)
Chills (General disorders) | 9 (11) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (11) | 10 (11)
Vomiting (General disorders) | 6 (7) | 7 (7)
Anorexia (General disorders) | 6 (6) | 4 (4)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Altered mental status (Psychiatric disorders) | 0 (0) | 1 (1)
Elevated ALT level (Hepatobiliary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No